CLINICAL TRIAL: NCT01118078
Title: Therapeutically Applicable Research to Generate Effective Treatments (TARGET) Initiative High-Risk Renal Tumor Project: Application of Array-Based Methods and Next Generation Sequencing to Identify Candidate Molecular Targets for High-Risk Wilms Tumors
Brief Title: Biomarkers in Tissue Samples From Patients With High-Risk Wilms Tumor
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AREN10B2; NCI-2011-02230 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000672402 (Other: Clinical Trials.gov); U10CA098543 (NIH); COG-AREN10B2 (Other: Children's Oncology Group)
Record Dates: First submitted 2010-05-05; First posted 2010-05-06 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Clear Cell Sarcoma of the Kidney; Recurrent Wilms Tumor and Other Childhood Kidney Tumors; Rhabdoid Tumor of the Kidney; Stage I Wilms Tumor; Stage II Wilms Tumor; Stage III Wilms Tumor; Stage IV Wilms Tumor; Stage V Wilms Tumor
MeSH Terms: conditions — Wilms Tumor | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis; Reverse Transcriptase Polymerase Chain Reaction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Archived tumor tissue samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Biomarker (DNA methylation, gene expression, RT-PCR): Archived tumor tissue samples are analyzed for DNA copy number determination, gene expression analysis, DNA methylation, and genomic re-sequencing by microarray analysis-based methods, including PCR analysis, DNA methylation analysis-specific RT-PCR, and quantitative RT-PCR (reverse transcriptase-polymerase chain reaction)
  Interventions: Genetic: DNA methylation analysis; Genetic: gene expression analysis; Genetic: microarray analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: diagnostic laboratory biomarker analysis

INTERVENTIONS:
Genetic: DNA methylation analysis — Undergo DNA methylation analysis
Genetic: gene expression analysis — Undergo gene expression analysis
Genetic: microarray analysis — Undergo microarray analysis
  Other Names: gene expression profiling
Genetic: reverse transcriptase-polymerase chain reaction — Undergo RT-PCR
  Other Names: RT-PCR
Other: diagnostic laboratory biomarker analysis — Correlative studies

SUMMARY:
This research study is studying biomarkers in tissue samples from patients with high-risk Wilms tumor. Studying samples of tissue from patients with cancer in the laboratory may help doctors to learn more about changes that occur in DNA and identify biomarkers related to cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To assess genomic gains and losses in high risk renal tumors, including up to 80 favorable histology Wilms tumors that relapse (RFHWT), 50 anaplastic Wilms tumors (UHWT), 15 clear cell sarcomas of the kidney (CCSK), and 40 rhabdoid tumors (RT) using a high density genetic platform to survey for recurrent copy number variations and allelic imbalances. II. To define transcription patterns within 80 RFHWT, 50 UHWT, 15 CCSK, and 40 RT using a high throughput platform for global gene expression. III. To define DNA methylation patterns within 80 RFHWT, 50 UHWT, 15 CCSK, and 40 RT using a high throughput platform. IV. To identify genetic mutations involved in the pathogenesis of Wilms tumor, and in the development of relapse and anaplasia through the study of 80 RFHWT, 50 UHWT, 15 CCSK, and 40 RT using next generation sequencing tools.

V. To facilitate the integration of the above databases and allow meaningful access by investigators through the infrastructure provided by TARGET, including its data portal and associated caBIG tool.

OUTLINE: This is a multicenter study.

Archived tumor tissue samples are analyzed for DNA copy number determination, gene expression, DNA methylation, and genomic re-sequencing by array-based methods, including PCR analysis, methylation-specific reverse transcriptase-PCR (RT-PCR), and quantitative RT-PCR.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high-risk Wilms tumor meeting ≥ 1 of the following criteria:

  * Relapsed disease
  * Anaplastic disease
  * Clear cell sarcomas of the kidney
  * Rhabdoid tumors
* Registered on NWTS-4, NWTS-5 (now COG-Q9401), or participation in AREN03B2 protocols with clinical follow-up > 3 years
* Banked frozen tumor samples and paired normal DNA available with clinical data points, including the following:

  * Age, race, and gender
  * Stage and reason for stage
  * Tumor weight
  * Associated precursor lesions (rests)
  * Histologic subtype
  * Site and time of recurrence
  * Days of follow-up
  * Time and reasons for death (e.g., tumor, toxicity, infection, or other)

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Up to 80 favorable histology Wilms tumors that relapse (RFHWT), 50 anaplastic Wilms tumors (UHWT), 15 clear cell sarcomas of the kidney (CCSK), and 40 rhabdoid tumors (RT)
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2010-05; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Genomic gains and losses in high-risk Wilms tumor | After completion of biomarker analysis
Transcription patterns involved in the pathogenesis of Wilms tumor | After completion of biomarker analysis
Genetic mutations involved in the pathogenesis of Wilms tumor | After completion of biomarker analysis

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Perlman, MD, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States